CLINICAL TRIAL: NCT06645067
Title: Cachectic Cancers and Adapted Physical Activity Assessment and Modulation of Energy Balance in Cachectic Patients Using Adapted Physical Activity
Brief Title: Assessment and Modulation of Energy Balance in Cachectic Patients Using Adapted Physical Activity
Acronym: EMC2APA
Status: Not yet recruiting | Type: Observational
Sponsor: University of Rennes 2 (Other)
Responsible Party: Principal Investigator, Peyrachon Romane, MD, University of Rennes 2
Other Study IDs: 2024-035
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Cancer Cachexia (CC); Exercise; Energy Regulation
Keywords: Cancer Cachexia; Exercise; Endurance; Energy Expenditure; Food Intake; Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cancer cachectic patients: This group is made up of patients suffering from cancer cachexia who take part in an APA programme at the medical-sports centre. These are patients who agree to have their energy expenditure measured at rest and during sub-maximal effort, as well as their level of physical activity and diet monitored for 7 days.
  Interventions: Behavioral: Measuring energy balance

INTERVENTIONS:
Behavioral: Measuring energy balance — The exercise intervention will consist of a personalized and supervised program lasting 12 weeks with two sessions per week, held on Tuesdays and Thursdays at the Sports and Medicine Center SPORMED in Rennes, France.
  Each session will combine endurance and resistance training, commencing with a 6-minute cardiovascular warm-up on ergometers (cycling ergometer or treadmill). This will be followed by 20 minutes at moderate intensity (60-70% of Heart Rate Reserve (HRR)), concluding with a 2-minute recovery period at light intensity. We will measure the resting ED at the start of the programme and the ED during moderate aerobic exercise in the 5th week of APA.

SUMMARY:
1. OBJECTIVE OF THE STUDY The study consists of evaluating resting energy expenditure (REE) and that induced by adapted physical activity (APA) in cachectic patients, compared with those predicted by equations and those of non-cachectic cancer patients. We will also seek to identify potential compensations in the level of Physical Activity (PA) and dietary intake during one week of the PA programme.
2. CONDUCT OF THE STUDY Taking part in this study will in no way affect your treatment at SPORMED; you will undergo the same assessments and carry out the PAA programme in the same way. As a reminder, your treatment at SPORMED consists of an initial assessment session, a 12-week ABS programme and a final assessment session.

If you take part in the EMC2APA study, we will ask you to measure your gas exchange at rest (60 minutes) and during the aerobic part of one of your physical activity sessions. You will perform the effort traditionally targeted during the sessions (constant moderate intensity (60% of your Reserve Heart Rate, equivalent to a perception of the difficulty of the effort of 5-6/10) while your gas exchanges will be measured using a portable, non-invasive measuring device (K5, COSMED®). You will also be fitted with an accelerometric wristwatch.

In addition to the gas exchange measurements that will take place in the SPORMED structure, we will ask you to fill in a logbook tracking your daily physical activity and your daily food intake. You will also be asked to wear an accelerometer in a belt attached to your hip for 7 days.

Participation in this study is voluntary. There are no restrictions during the protocol.

DETAILED DESCRIPTION:
To stabilize patients' weight, it is essential to measure energy expenditure in order to propose appropriate nutritional and physical activity management (Purcell et al., 2016; Vazeille et al., 2017; Barcellos et al., 2021). In clinical practice, nutritional management is often based on predictive equations for end-stage renal disease (ESRD). These predictive equations include parameters such as age, height, weight, and sex. The most widely used is the Harris and Benedict equation, in which 85% of the healthy population has a resting energy expenditure (REE) between 90 and 110% of the predicted value. However, Barcellos et al. (2021) demonstrate that this equation underestimates REE by 648 kcal/day compared to values measured by indirect calorimetry in cancer patients. Predictive equations, therefore, seem obsolete for cancer patients, despite the central role of energy balance in treatment.

Several factors reduce the relevance of these equations and highlight the need for specific measurement of REE and total energy expenditure (TEE). Tumor type, size, and stage influence energy expenditure (Tuccar et al., 2021). A meta-analysis by Nguyen et al. (2016), including 27 studies, shows that REE increases by 9.66 kJ/kg fat-free mass (FFM)/day in cancer patients. REE can increase from 100 to 1400 kcal/day depending on tumor type (Purcell et al., 2016). However, tumor type directs the magnitude and direction of changes in energy metabolism. In a review by Hanna et al. (2023), the lean mass-adjusted REE shows that patients with high gastrointestinal cancers have higher REE than healthy individuals in 6 of the 9 studies, while the other 3 studies reported similar REE (Hanna et al., 2023). Tumors of the lung, head and neck, esophagus, stomach, liver, and pancreas are most affected by hypermetabolism (REE > 110% of predicted values), whereas melanoma, colorectal, and breast cancers show more normal metabolism (90 < REE < 110% of predicted values) or even hypometabolism (REE < 90% of predicted values) (Dempsey et al., 1984; Hanna et al., 2023; Tuccar et al., 2021; Purcell et al., 2016).

Determining the energy expenditure induced by physical activity (PA) in the presence of cachexia would allow for better nutritional management and contribute to further understanding of cancer cachexia management. Moreover, objectively assessing the different components of total energy expenditure (TEE), such as activity energy expenditure (AEE), would validate or challenge the use of predictive equations based on healthy individuals, identifying the specific needs of cachectic patients in terms of TEE and AEE induced by PA. Objective measurement of AEE will be more reliable than subjective estimates using questionnaires, which are prone to over- and under-estimation biases (Purcell et al., 2019). Altogether, this will enable more precise nutritional and PA recommendations for patients.

Objectives

The study aims to evaluate resting energy expenditure (REE) and PA-induced expenditure in cachectic patients compared to values predicted by equations and those in non-cachectic patients. The goal is also to assess potential compensatory effects on PA levels and daily intake during PA sessions.

General Hypotheses

Based on the literature, cachectic patients are expected to exhibit hypermetabolism, with REE values ≥ 110% of the values predicted by equations. Additionally, REE expressed as kcal/day/kg of lean body mass is expected to be higher in cachectic patients compared to non-cachectic patients due to chronic inflammation and tumor-related energy expenditure.

Regarding AEE, no studies have focused on this parameter in cachectic patients. TEE is mostly estimated using approximate predictive equations, with only one study by Moses et al. (2004) addressing TEE in cachectic patients. This study aims to characterize energy expenditure induced by moderate-intensity exercise to adjust nutritional interventions according to patients' PA levels.

Regarding daily PA levels, it is hypothesized that cachectic patients reduce daily PA on PA session days to compensate for energy expenditure (Moses et al., 2004). Additionally, individuals are expected to increase their food intake to maintain energy balance and benefit from symptom reduction provided by PA.

Assessment of Resting and Exercise Energy Expenditure: REE and exercise energy expenditure (EEE) measurements are standardized at the SPORMED facility. If consent is obtained (Consent form in the appendix), data may be transferred to a secure data collection file for analysis. Data will be stored on an external password-protected hard drive and on the Huma-Num University data management server.

Assessment of Eating and Physical Activity Behaviors: Dietary behavior will be monitored over a 7-day period using a nutrition diary. PA behavior (duration and intensity, including vigorous, moderate, light activity, walking, sedentary behavior, and sleep duration) will be measured using a validated accelerometer (wGT3X+) worn at the hip. If consent is obtained, data will be transferred to a data collection file for analysis. Handwritten dietary data will be digitized, and accelerometer data will be extracted. All data will be securely stored.

Variables and Measurement Tools:

Assessment of Resting and Exercise Energy Expenditure: Using the K5 (COSMED®), a portable, non-invasive metabolic system for field and lab tests.

Resting Energy Expenditure (REE): Patients will avoid moderate and vigorous PA for 24 hours before the measurement, as well as a 4-hour fast. No caffeine is allowed for 4 hours and no tobacco for 2.5 hours. During the measurement, patients will rest in a lying position for 30 minutes. The measurement lasts 10 minutes once a stable state is reached (oxygen consumption varies by less than 10%) (Rey, 2018). The room temperature will be kept between 22 and 25°C to limit environmental effects on energy expenditure (Fullmer et al., 2015).

Exercise Energy Expenditure (EEE): Conducted on a treadmill or stationary bike, the measurement includes a 7-minute warm-up, with incremental intensity to reach moderate effort (RPE 5/10 or 60% of max HR), followed by 15 minutes of constant effort. A 2-minute recovery will be included. The data collected will help assess respiratory function and estimate energy expenditure using the Weir equation.

Heart rate, subjective effort perception, and PA "counts" will also be recorded to compare energy expenditure estimates from predictive equations and activity monitors. Dietary intake and appetite will be recorded daily in a nutrition journal, with a 7-day monitoring period.

Study Duration: The number of subjects required was based on Moses et al.'s (2004) study. An estimated 5 patients per group are needed, considering REE and EEE, with a study duration of 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old.
* Have understood the objectives of the study.
* Have read and signed the consent form.
* Be affiliated with a social security system.
* Currently undergoing cancer treatment.

Exclusion Criteria:

* Une fatigue extrême
* Une anémie symptomatique (hémoglobine ≤ 8 g/dl)
* Un syndrome infectieux sévère en cours d'évolution
* Une décompensation de pathologie cardio-pulmonaire
* La présence de lésions osseuses lytiques du rachis ou des os longs (la contre-indication concerne la mobilisation du membre atteint)
* Une intolérance au port du masque de l'appareil K5 (Cosmed)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cachectic cancer patients: patients who have lost weight significantly in the last 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Exercise energy expenditure | During an exercise session in the 5th week of the programme.
  The measurement will be carried out on a treadmill ergometer and/or stationary bike. The exercise energy expenditure measurement will include a 7-minute warm-up with incremental intensity to reach a work level representing moderate effort in terms of RPE (5/10) or heart rate (60% of maximum heart rate), followed by 15 minutes of constant moderate-intensity exercise. A 2-minute recovery period will be added at the end to avoid abrupt physiological changes. The exercise energy expenditure measurement will take place after a period of familiarization with the cycle ergometer to minimize disturbances caused by stress or technical inefficiency.

SECONDARY OUTCOMES:
Resting Energy Expenditure | During the initial consultation before starting the exercise programme
  Patients will be instructed to avoid moderate and vigorous physical activities for 24 hours prior to the measurement. Additionally, a 4-hour fast will be required, with no caffeine consumption during the last 4 hours and no tobacco use during the last 2.5 hours. During the measurement, patients will lie down for 30 minutes to reduce energy expenditure from previous physical activity. The measurement will then last 10 minutes once a stable state is reached (period during which oxygen consumption varies by less than 10%) (Rey, 2018). The room temperature will be maintained between 22 and 25°C to limit the effects of a cold environment on energy expenditure (Fullmer et al., 2015).
Physical Behavior : Moderate Physical Activity | Over 8 days during the exercise program
  Moderate physical activity will be evaluated using the Steel HR (Withings®) activity monitors and the wGT3X+/GT3X+ accelerometers (ActiGraph®) worn at the waist (Smith et al., 2020), as well as a logbook documenting physical activities lasting longer than 10 minutes.
Dietary Intake and Appetite | For 8 days during the exercise program
  Dietary intake and appetite will be recorded daily in a nutrition journal, which is the reference method (Ortega et al., 2015), and using the SEFI® scale (Simple Evaluation of Food Intake) (Thibault et al., 2021). We will ensure a period of familiarization with the tool before the 7-day measurement period. The journal will allow us to assess appetite perception, meal frequency, quantities consumed, and any potential disruptions. These elements will help identify possible variations related to the completion of APA sessions.
Subjective Effort Perception | During Exercise Energy Expenditure assessment
  Subjective effort perception (RPE) will be assessed using the modified Borg scale ranging from 1 to 10. This scale helps to subjectively assess effort intensity, especially since certain antitumor treatments can alter heart rate responses to exercise.
Heart Rate | During Exercise Energy Expenditure assessment
  During both energy expenditure measurements with the K5 (COSMED®), heart rate (HR) will also be measured using a heart rate monitor.
Physical behavior : Vigorous Physical activity | Over 8 days during the exercise program
  Vigorous physical activity will be evaluated using the Steel HR (Withings®) activity monitors and the wGT3X+/GT3X+ accelerometers (ActiGraph®) worn at the waist (Smith et al., 2020), as well as a logbook documenting physical activities lasting longer than 10 minutes.
Physical behavior : Walking duration | Over 8 days during the exercise program
  Walking duration will be evaluated using the Steel HR (Withings®) activity monitors and the wGT3X+/GT3X+ accelerometers (ActiGraph®) worn at the waist (Smith et al., 2020), as well as a logbook documenting walking activities lasting longer than 10 minutes.
Physical Behavior : Sitting time | Over 8 days during the exercise program
  Sitting time will be evaluated using the Steel HR (Withings®) activity monitors and the wGT3X+/GT3X+ accelerometers (ActiGraph®) worn at the waist (Smith et al., 2020).
Physical Activity Counts | During Exercise Energy Expenditure assessment
  During both energy expenditure measurements with the K5 (COSMED®) physical activity "counts" will also be measured using a wrist-worn accelerometer. This data will allow comparison of energy expenditure estimates derived from predictive equations and activity monitors (smartwatches).
Daily Physical Activity Counts | For 8 days during the exercise program
  Daily physical activity "counts" will be measured with the wGT3X+/GT3X+ accelerometers (ActiGraph®). This data will allow comparison of energy expenditure estimates derived from predictive equations and activity monitors (smartwatches).

CONTACTS AND LOCATIONS:
Locations (1):
- SPORMED, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: Undecided